CLINICAL TRIAL: NCT07048600
Title: A Pilot Randomized Trial of Brief Standalone Group Acceptance and Commitment Therapy (ACT-i) for Chronic Insomnia
Brief Title: Brief Trial of ACT-i for Adults With Chronic Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Roxana Cardos, Lect. Univ. Dr., Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 407/25.04.2025
Record Dates: First submitted 2025-05-20; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Chronic Insomnia; Depression - Major Depressive Disorder; Anxiety
Keywords: acceptance and commitment therapy; chronic insomnia; cognitive functions; depression; anxiety; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The main investigator and statistician of the study will be blinded to the randomization schedule, as a third party will perform the randomization and assign participants to the treatment groups. The online platform will generate the allocation after the inclusion and exclusion criteria are met and the pre-test forms are performed. Participants will be blind to their group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy for Insomnia (ACT-i) (Experimental): The intervention is available in its individual and group format, which can be adapted to an online context in "Acceptance and Commitment Therapy for Insomnia: A Session-By-Session Guide", by Renatha El Rafihi-Ferreira (Rafihi-Ferreira, 2024). It comprises the details of each ACT-i group session with illustrations and examples for the trained therapists.
  Participants will be requested to register to an Online Platform, such as Google Meet, to attend the two sessions which will be guided by a trained therapists. Each session will have approximately 120 minutes. They will receive instructions from the therapists and handouts at the end of each session. Facilitators will receive training from a specialized mental health professional.
  Interventions: Behavioral: Acceptance and Commitment Therapy for Insomnia
- Attentional Control Group (Active Comparator): Participants will receive this intervention in an online platform by a trained professional. His training will be provided by a mental health expert with experience in carrying out psychoeducational and non-directive group sessions. This group will match the ACT-i intervention in terms of session duration, delivery format, group interaction, facilitator contact, time and handouts/ homework.
  Interventions: Behavioral: Attentional Control Group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for Insomnia — Monotherapy ACT-i, with no behavioral components, is a brief and low-intensity treatment that has recently been detailed by experts in the field in a session-by-session guideline, intending to help people affected by chronic insomnia. The key components of the sessions are psychoeducation, mindfulness, values and actions derived from chosen values, and defusion.
  An adapted, brief and online version of the intervention was developed by the authors of this study. Both interventions were matched in terms of overall duration and delivery format. Each session was tailored to follow a comparable format. Therapeutic alliance, psychoeducation, sleep hygiene, relaxation training and homework was targeted in the first session. In the second session, ACT-i focused on values, acceptance strategies and psychological flexibility. This version will be published online upon request. Each session will last 120 min. They will be delivered once per week, for two consecutive weeks.
  Arms: Acceptance and Commitment Therapy for Insomnia (ACT-i)
Behavioral: Attentional Control Group — The focus of the sessions will be on participants, on general topics. It will not include any active, psychological intervention components, such as cognitive restructuring or ACT processes. No recommendations or psychological guidance will be given. Each session will last 120 minutes. It will be held once per week, for two weeks.
  Arms: Attentional Control Group

SUMMARY:
This is a prospective, randomized-controlled trial that assesses the efficacy of a brief Acceptance and Commitment Therapy (ACT-i), compared to an attentional control group, in adults with chronic insomnia. The interventions will be evaluated for their impact on insomnia severity, cognitive function, depression, anxiety, psychological flexibility, and sleep beliefs - measured before treatment, two weeks after and at a three-month follow-up.

DETAILED DESCRIPTION:
Insomnia is the most prevalent sleep disorder. It is associated with impairments both physically and psychologically. Therefore, it usually causes a suite of durable stressors in numerous aspects of life, such as academically, professionally, socially, and financially. Given its widespread impact, early effective treatments are crucial to prevent long-term consequences.

The first line of treatment is Cognitive-Behavioral Therapy for Insomnia (CBT-i). Despite its effectiveness, approximately 60% of individuals with chronic insomnia and comorbidities do not go into remission after treatment or simply do not adhere to it. Acceptance and Commitment Therapy for Insomnia (ACT-i) has great potential for overcoming this limitation, as it focuses on accepting the feelings and thoughts associated with insomnia, through value-based actions. However, more studies on ACT-i as a monotherapy are needed.

This study aims to evaluate the efficacy of brief, group ACT-i for chronic insomnia in adults, versus an attentional control group. Participants will be aged between 18 and 59 years, diagnosed with chronic insomnia who will be randomly assigned to either ACT-i, or the control group. To limit age-related sleep changes, only participants aged up to 59 will be included, as sleep difficulties tend to increase after the age of 60. The interventions will be performed in groups, in 2 weekly sessions. Their effects will be investigated for the primary outcome related to the severity of insomnia, and secondary outcomes related to depression, anxiety, cognitive functioning, psychological flexibility, and beliefs about sleep at pre-test, post-test at two weeks and three-month follow-up. After the interventions, participants will complete an inventory regarding the adherence and satisfaction to both interventions. This is the first attempt to investigate a group-based ACT-i as monotherapy with an attentional control group delivered in an accessible, brief-group format. Specifically, the sessions are implemented briefly in 2 group sessions, unlike other studies that have (at least) 4 group sessions. Furthermore, the investigators will also compare their adherence rates and patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* clinical/ subclinical diagnosis of chronic insomnia either already diagnosed by a professional, or identified with SCISD-R by our team of clinicians
* age over 18 and older, but not over 59 years old;
* minimal/ mild symptomatology of depression (scores ≤ 9 on PHQ-9) and/ or anxiety (scores ≤ 9 on GAD-7) or as diagnosed with SCID-5-CV;

Exclusion Criteria:

* diagnosed with a neurological degenerative disorder, or any moderate/ severe psychiatric disorder;
* diagnosed with other sleep disorder (e.g., sleep apnea, restless legs/ periodic limb movements, circadian-based sleep disorder);
* diagnosed with cognitive impairments;
* unable to understand Romanian;
* unable to attend to online-sessions (e.g., no laptop, microphone, camera);

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in the score of Insomnia Severity Index (ISI); | baseline, 2 weeks after the intervention
  The Insomnia Severity Index (ISI) is a brief tool of chronic insomnia. It consists of 7 items about the severity of insomnia, its noticeability, and daytime functioning. Total scores range from 0 to 28, with higher scores reflecting more severe clinical insomnia.

SECONDARY OUTCOMES:
Change in the score of Insomnia Severity Index (ISI) | 3 months after the intervention
  Follow-up evaluation of the severity of insomnia using ISI
Change in the score of Patient Health Questionnaire-9 | 3 months after the intervention
  The Patient Health Questionnaire-9 (PHQ-9) is a brief tool of depression. It consists of 9 items about depressive symptomatology, such as anhedonia, sadness and fatigue. Total scores range from 0 to 27.
Change in the score of Multidimensional psychological flexibility inventory (MPFI-24; Gregoire et al., 2020) | 3 months after the intervention
  The Multidimensional psychological flexibility inventory (MPFI-24) is a 24-item measure of psychological flexibility, including acceptance, mindfulness, and values-based actions. Total scores range from 24 to 144.
Change in the score of the Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) | 3 months after the intervention
  The Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) is a 16-item scale measuring dysfunctional sleep-related cognitions. Total score is added up and divided by 16, and a higher score represents higher unrealistic expectations regarding sleep.
Change in the score of The Cognitive Failures Questionnaire (CFQ) | 3 months after the intervention
  The Cognitive Failures Questionnaire (CFQ) is a self-report tool of the frequency of daily cognitive failures, such as forgetfulness or lapses in attention. It has 25 items and total scores range from 0 to 100, with higher scores indicating more subjective cognitive failure.
Change in the score of Barkley Deficits in Executive Functioning Scale (BDEFS-SF) | 3 months after the intervention
  The Barkley Deficits in Executive Functioning Scale (BDEFS-SF) is a 20-item self-report measure of executive functioning deficits. Each item is rated on a 4-point Likert scale, ranging from 1 ("never or rarely") to 4 ("very often"). Total scores range from 20 to 80.

OTHER OUTCOMES:
Satisfaction: Client Satisfaction Questionnaire (CSQ-8) | one day after the intervention
  The Client Satisfaction Questionnaire (CSQ-8) is a brief tool of general satisfaction with the treatment being given. Each item is rated on a 4-point scale, ranging from 1 ("weak") to 4 ("excellent"). Total scores range from 8 to 32, with higher scores reflecting greater satisfaction.
Adherence: Adherence and satisfaction questionnaire (Ferreira et al., 2024) | one day after the intervention
  Adherence and satisfaction questionnaire is a brief self-report tool of adherence and satisfaction with the provided treatment. It has 8 items, with yes and no answers.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
Will share IPD used in the results of the publication, upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD may be shared after publication upon request, with no end date.